CLINICAL TRIAL: NCT06264466
Title: Safety and Efficacy of the Novel Speedboat UltraSlim With Radiofrequency and Microwave Ablation Flexible Biplolar for Per-Oral Endoscopic Myotomy in Patients With Achalasia: A Single Center Prospective Study
Brief Title: Safety and Efficacy of a Novel Flexible Bipolar in POEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IECED-010112023
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Esophageal Achalasia
Keywords: achalasia; POEM; Radiofrequency; microwave
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: interventional trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POEM with Speedboat Ultraslim (Experimental): Participants aged 18-years and above, referred to the participating center (IECED) with a diagnosis of achalasia and indication for POEM, POEM procedures will be performed using the Speedboat UltraSlim
  Interventions: Device: POEM with Speedboat Ultraslim

INTERVENTIONS:
Device: POEM with Speedboat Ultraslim — POEM procedures, with or without fundoplication, will be conducted by expert endoscopists who have undergone prior training in the utilization of the ultraslim Speedboat. Incisions, whether anterior or posterior, submucosal tunneling, and myotomy will be performed using the Bipolar Radiofrequency Ablation (RFA) integrated into the device's tip. Additionally, for vessel coagulation, the microwave energy integrated into the device's tip will be employed. Successful myotomy will be confirmed by passage of the endoscope through the esophagogastric junction (EGJ) without restriction.

SUMMARY:
Per-oral endoscopic myotomy (POEM) is a minimally invasive therapy for achalasia. The procedure has demonstrated high technical and clinical success with lower adverse events. Different types of knives have been used for cutting and coagulation during the procedure; however, exchanging accessories is sometimes needed to perform all the stages of POEM.

To overcome this disadvantage, the investigators aim to evaluate a single device that integrates in its tip bipolar radiofrequency and microwave, the Speedboat Ultraslim (Creo Medical, UK) for cutting and coagulation during POEM procedure. Some of the promise's advantages derived from its use are: (1) less inflammation, (2) clear differentiation between layers, (3) the use of a single device for the procedure.

This single-center, prospective, interventional study will include patients with achalasia submitted to POEM procedure, with or without fundoplication (POEM-F). All stages (mucosal incision, submucosal tunneling, myotomy) of POEM will be performed using the Speedboat ultraslim flexible catheter. Technical and clinical success, along with safety will be the primary endpoints; while, post-procedure reflux symptoms and quality of life will be assessed as secondary outcomes with reflux severity index (RSI) and the Northwestern Esophageal Quality of Life (NEQOL), respectively.

DETAILED DESCRIPTION:
Achalasia is characterized by the absence of esophageal peristalsis and the inability of the lower esophageal sphincter (LES) to relax. To date, the therapies with higher success rates are the Heller myotomy and the minimally invasive per-oral endoscopic myotomy (POEM). Different tools have been developed for the different POEM stages (mucosal incision, submucosal tunneling, myotomy, and closure). However, some devices need exchanging accessories for cutting and coagulation.

In light of the above, the investigators aim to evaluate a newly launched ultra-slim flexible catheter, Speedboat Ultraslim (Creo Medical, UK) that integrates bipolar radiofrequency (RFA) energy and microwave in its tip for cutting and coagulation, respectively, in patients with achalasia. Some proposed advantages of using this device during POEM are (1) less inflammation and better healing process derived from localized bipolar energy; (2) a protective full that facilities clear differentiation between muscular and mucosal layers; (3) the use of a single device to complete the POEM procedure.

After completing the inclusion criteria, the patients with achalasia will undergo POEM (anterior or posterior incision) with or without fundoplication (F-POEM). The procedures will be performed by previously trained expert endoscopist. The mucosal incision, submucosal tunneling and cutting will be performed using RFA energy, while coagulation will be performed with microwave, both integrated in the tip of the Ultraslim Speedboat.

Technical and clinical success along with safety will be the primary outcomes; while post-procedure reflux symptoms and quality of life will be assessed as secondary outcomes with reflux severity index (RSI) along with endoscopic and pH studies; and the Northwestern Esophageal Quality of Life (NEQOL), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years of age or older.
* Patients referred to the participating center (IECED) with a clinical diagnosis of achalasia with an indication for POEM, including previously failed Heller myotomy, balloon dilation or POEM
* Patients who provide informed consent.

Exclusion Criteria:

* Patients who have contraindications for esophagogastroduodenoscopy (EGD).
* Patients with an Eckardt score < 3 before POEM.
* Positive diagnosis of Chagas disease.
* Patients unable to withstand general anesthesia.
* Pregnancy and lactation.
* Barret's esophagus.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Technical success of procedure | up tp four hours
  Successful competition of all the stages of the POEM procedure with passage of endoscope through the EGJ.
Clinical success of procedure | up to one year
  The clinical success of the POEM procedure will be assessed by using the Eckardt score. An Eckardt score of ≤3 will be considered as clinical success.
Frequency of adverse events attributable to the procedure | Up to three months
  Frequency of adverse events attributable to the procedure, based on American Society of Gastrointestinal Endoscopy (ASGE) lexicon.

SECONDARY OUTCOMES:
Rate of Gastroesophageal reflux disease | Up to one year
  The diagnosis of gastroesophageal reflux disease will be based in one or more of the following criteria:
  1. Endoscopic Erosive Esophagitis, LA grade B or above
  2. Long segment Barrett´s esophagus
  3. Peptic esophageal stricture
  4. 24-hour pH study with acid exposure time >6%
  For endoscopic and pH study, proton pump inhibitors should be stopped for two to four weeks.
Assessment of Gastroesophageal reflux disease severity | Up to one year
  The gastroesophageal reflux will be clinically assessed by the reflux symptoms index (RSI). The RSI consists in nine items that assess various symptoms related to GERD. RSI ≥13 related to significant reflux disease.
Change in health-related quality of life after POEM | Up to six months
  Effect in the Gastroesophageal reflux disease health-related quality of life through the Northwestern Esophageal Quality of Life (NEQOL) scale.
  NEQOL, a 14-item, single-scale measure of Health-related quality of life (HRQOL), that allows for rapid assessment in a clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas (IECED)
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas (IECED), Guayaquil, Guayas, Ecuador

REFERENCES:
- [Background] Rolland S, Paterson W, Bechara R. Achalasia: Current therapeutic options. Neurogastroenterol Motil. 2023 Jan;35(1):e14459. doi: 10.1111/nmo.14459. Epub 2022 Sep 25. PMID 36153803
- [Background] Tasnim S, Raja S, Sudarshan M. Achalasia: Surgery Versus Per-Oral Endoscopic Myotomy. Thorac Surg Clin. 2023 May;33(2):135-140. doi: 10.1016/j.thorsurg.2023.01.007. Epub 2023 Feb 26. PMID 37045482
- [Background] Patil G, Dalal A, Maydeo AP. Feasibility of Speedboat RS2 with bipolar radiofrequency energy for peroral endoscopic myotomy in patients with achalasia (with video). Endosc Int Open. 2020 Aug;8(8):E998-E1001. doi: 10.1055/a-1165-0087. Epub 2020 Jul 21. PMID 32743048